CLINICAL TRIAL: NCT06739096
Title: Investigation of the Effectiveness of Short Wave Diathermy Treatment in Patients With Hand Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Sezgin (Other)
Responsible Party: Sponsor-Investigator, Omer Sezgin, MD, Haydarpasa Numune Training and Research Hospital
Organization: Haydarpasa Numune Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HNHEAH-KAEK 2024/36
Record Dates: First submitted 2024-12-08; First posted 2024-12-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-12

CONDITIONS: Hand Osteoarthritis; Osteoarthritis
Keywords: hand osteoarthritis; short wave diathermy; shortwave diathermy
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short Wave Diathermy + Exercise (Experimental)
  Interventions: Device: Short Wave Diathermy; Other: Exercise
- Sham Short Wave Diathermy + Exercise (Sham Comparator)
  Interventions: Other: Exercise; Device: Sham Short Wave Diathermy

INTERVENTIONS:
Device: Short Wave Diathermy — Shortwave diathermy (SWT) is a form of electromagnetic therapy that causes the movement of ions, the disruption of molecules, and the generation of eddy currents, which ultimately produce heat in deep tissue. Its claimed mechanism of action includes inducing an anti-inflammatory response, reducing joint stiffness, stimulating connective tissue repair, and reducing muscle spasm and pain.
  Arms: Short Wave Diathermy + Exercise
Other: Exercise — range of motion, strengthening and stretching exercises
Device: Sham Short Wave Diathermy — Sham protocol
  Arms: Sham Short Wave Diathermy + Exercise

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled study was to evaluate the effects of shortwave diathermy therapy on pain, grip strength, and functionality in patients with hand osteoarthritis.

DETAILED DESCRIPTION:
Patients who apply to the physical medicine and rehabilitation outpatient clinic between January 2024 and February 2025 will be included in the study according to the inclusion and exclusion criteria specified below. Demographic data of the patients such as age, gender, height, and weight will be recorded. In the initial evaluation, VAS, hand dynamometer and pinchmeter measurements, Duruöz Hand Index questionnaire and Moberg Addition Test results of the patients will be noted. The G*Power 3.1 (Faul, Erdfelder, Lang, and Buchner, 2007) program was used to calculate the sample size. In the comparisons of different parameters between groups in reference studies, the effect size was calculated to be at the level of 0.9. This corresponds to a large level according to Cohen's effect size classification. Accepting a statistical significance coefficient of 0.05 with an effect size of 0.9, it was decided to include a minimum of 16 people in each group to obtain 80% power. A total of 36 patients (with a 10% drop-out margin) will be included in the study and will be randomly divided into two groups as treatment and control groups. Randomization will be done by closed envelope method. The treatment group will be given 15 sessions: 20 minutes (27.12 MHz, continuous mode, 400W output) short wave diathermy treatment, hand osteoarthritis exercise program. The control group will be given 15 sessions: sham short wave diathermy and hand osteoarthritis exercise program. Patients will complete 15 sessions, 1 session per day, 5 sessions per week. All evaluation parameters will be recorded before treatment, at the end of treatment and at the end of treatment at the 12th week. Intra-group and inter-group differences will be examined statistically.

ELIGIBILITY:
Inclusion Criteria:

* To be between 35-75 years old
* Diagnosis of hand osteoarthritis according to the ACR 1990 Criteria

Exclusion Criteria:

* Chronic inflammatory diseases (rheumatoid arthritis, seronegative spondyloarthropathy, gout, hemochramatosis, etc.)
* Malignancy
* Having uncontrolled systemic disease (cardiovascular, pulmonary, hematologic, hepatic, renal, endocrinologic)
* Synovitis, tenosynovitis, entrapment neuropathy, contracture, open wound in hand/wrist
* History of hand fracture and/or operation
* Regular use of nonsteroidal anti-inflammatory drugs in the last three weeks
* Regular use of diaserin, chondroitin sulfate, glucosamine in the last three months
* Body Mass Index greater than 35

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | At the beginning of treatment (week 0), at the end of treatment (week 3) and 12 weeks after the end of treatment (week 15)
  0-10 scale. Higher scores represent more severe pain.
hand dynamometer and pinchmeter measurements | At the beginning of treatment (week 0), at the end of treatment (week 3) and 12 weeks after the end of treatment (week 15)
  Measurements will be made three times for each fine force on both hands and the average values will be recorded in kg.

SECONDARY OUTCOMES:
Duruöz Hand Index | At the beginning of treatment (week 0), at the end of treatment (week 3) and 12 weeks after the end of treatment (week 15)
  It is a self-report functional disability scale containing 18 items on daily living activities. Each question is scoring from 0 to 5. The total score ranges from 0 to 90. A higher score indicates a greater level of limitations.
Moberg Pickup Test | At the beginning of treatment (week 0), at the end of treatment (week 3) and 12 weeks after the end of treatment (week 15)
  In the Moberg pick-up test, for the evaluation of hand skills, the patient was positioned in the sitting position in a chair and a table was put in front of the patient, and 8 small objects were put on the table . The patient was requested to pick up these objects using the affected hand without sliding on the surface and to put them in a box present on the table, and the duration was recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Mesci, Assoc. Prof., MD, Study Chair — Haydarpaşa Numune Training and Research Hospital; Duygu Geler Külcü, Prof., MD, Study Director — Haydarpaşa Numune Training and Research Hospital; Sibel Süzen Özbayrak, MD, Study Director — Haydarpaşa Numune Training and Research Hospital
Locations (1):
- Haydarpaşa Numune Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Safety concerns